| Protoni | cs Knee | Brace | versus | Hamstring | Resisted | Exercise | (HRE) |
|---|---|---|---|---|---|---|---|
| | on Indiv | viduals | With Pa | atellofemo | ral Pain Sy | yndrome | |

01/11/2017

NCT03042559

IRB #: 5160417

# Methodology

# Design

This study is a randomized controlled trial with two treatment groups – the Protonics<sup>TM</sup> knee brace group and the sport cord group. Subjects with PFPS were asked to complete a series of open-chain hamstring resistance exercises with either apparatus, for which the procedures are described below, for four weeks. After the intervention, knee joint function and clinical symptoms of PFPS were assessed and compared between groups.

## **Participants**

Subjects were recruited based on the following inclusion criteria: male or female 18-45 years of age; has exhibited patellofemoral pain symptoms for more than 1 month and have a pain level  $\geq 3$  on the NPRS; has experienced pain during at least 2 functional activities, such as squatting, ascending/descending stairs, and/or running. Individuals who had experienced traumatic injuries to the knee joint or lower extremity, displayed signs or symptoms of a meniscus lesion or ligamentous-related pathology, had been diagnosed with a neurological disorder, diabetes, osteoarthritis, osteoporosis, or rheumatoid arthritis, or reported taking any over-the-counter pain medications during the study period were excluded from the study. Screening of subjects was done by a licensed physical therapist under the supervision of an Orthopedic Clinical Specialist (OCS) with over 29 years of experience.

Flyers, emails, phone calls, and referrals were used to gather a convenience sample of subjects. Subjects were randomly assigned to either the Protonics<sup>TM</sup> knee brace group or the sport cord group using simple randomization (Figure 1). All participants were required to sign an informed consent form. This study was approved by the Loma Linda University Institutional Review Board and was registered at http://clinicaltrials.gov (registration number NCT03042559).

### **Procedures**

Subjects assigned to the Protonics<sup>TM</sup> knee brace group were asked to perform warm up exercises, followed by specific therapeutic exercises that are part of the Protonic Therapy Program (PTP)<sup>18</sup>. The Protonics system has been introduced to physical therapists as a potential treatment for PFPS. The system includes a brace set to resist knee flexion and a set of specific exercises to perform daily. Through resistance to knee flexion, the system is advertised to decrease retropatellar contact pressure due to changes in pelvis inclination and available hip rotation. Specifically, resistance to knee flexion is purported to increase hamstring activity and inhibit the activity of the tensor fasciae latae and psoas muscles. The manufacturer asserts that prolonged use of the system results in greater hamstring activation, which leads to permanent structural changes through reciprocal inhibition at the hip and pelvis<sup>18</sup>. The phases of the intervention are summarized in Table 1. The warm-up consisted of the subject wearing the Protonics<sup>TM</sup> knee brace set at a moderate resistance level and flexing the knees while sitting, standing, and reclining in the supine and prone positions. The exercises, were done in sets of 10-15 repetitions, 3 sets per day, 3 times per week, for 4 weeks. Each set took about 5 minutes for subjects to complete, or 15 minutes per day.

The PTP has three phases. At the start of each phase, subjects were given detailed instructions on how to perform the warm up and therapeutic exercises and instructed to perform them at home 3 times per week. During Phase I or day 1, subjects were asked to walk for 5 minutes or as tolerated at varying speeds while wearing the brace. Subjects also performed the Protonics<sup>TM</sup> gait and Protonics<sup>TM</sup> neuromuscular repositioning techniques. During Phase II or weeks 1 and 2, subjects performed the same Protonics<sup>TM</sup> techniques, and were asked to walk for 8 minutes or as tolerated at varying speeds and inclines. Subjects were also instructed to perform 10-15 repetitions of the hamstring curl in the prone, supine, and seated positions at home. The seated hamstring curl

is displayed in Figure 2. During Phase III or weeks 3 and 4, subjects were once again asked to perform the aforementioned Protonics<sup>TM</sup> techniques, but this time they were also asked to walk forwards and backwards at varying speeds and inclines for 10 minutes or as tolerated. They were also instructed to do 10-15 repetitions of the standing hamstring curl.

Subjects assigned to the sport cord group were asked to do the same warm-ups and exercises using the sport cord in the supine, standing, sitting, and prone positions. The prone hamstring curl can be seen in Figure 3. The only difference is that subjects were asked to only walk backwards instead of forwards in order to avoid activation of the hip flexor muscle. The appropriate level of resistance for each subject was calculated by multiplying their weight in pounds by 0.3. Subjects were then given either light, medium, or heavy resistance cords according to the following classification scheme: light (pink color) with resistance 3 (R3), 0-30 lbs.; medium (orange color) with resistance 5 (R5) 0-50 lbs.; heavy (yellow color) with resistance 7 (R7) 0-70 lbs. All subjects completed three study visits, and a total of four measurements were taken at baseline, immediately following the first session, at two weeks, and at 4 weeks.

# **Compliance**

Several methods were employed to maximize subjects' compliance: During the initial visit, subjects were provided a thorough educational session on the appropriate use of the sport cord and knee brace and were given the opportunity to ask questions at any point of the study. The educational session included oral instructions as well as brochures which subjects could refer to for complete written instructions and visual depictions of the prescribed exercises. As the study was divided into three phases, subjects were asked to visit the lab at least three times and to return for additional visits if they wished. Additionally, a log sheet was filled out by each subject to track

completion of his/her exercises at home. Finally, text message reminders were sent to each subject throughout the study.

#### **Outcome Measures**

The primary outcome measures of the study can be divided into two categories: clinical outcomes and functional outcomes.

#### Clinical Outcome Measures:

APT was assessed using a palpation meter (PALM) inclinometer with the subject in the standing position; one arm of the caliper was placed on the anterior superior iliac spine (ASIS) while the other was positioned on the posterior superior iliac spine (PSIS). This technique was shown to be a reliable way of assessing sagittal pelvic position <sup>19</sup>. As described by Herrington, subjects were required to stand on a 30 centimeter high platform, look forward at a fixed point, and keep their arms crossed over their chest during palpation <sup>20</sup>.

Hip internal/external rotation active range of motion (ROM) was measured from sitting position as follows: the measured hip was placed at 90 degrees flexion, in neutral position between adduction and abduction, and knee joint at 90 degrees flexion, as described by Han and colleagues <sup>21</sup>. While the contralateral hip placed on 30 degrees abduction. Using a fluid-filled inclinometer placed parallel to the shaft of distal tibia and proximal to medial malleolus. The tibia was vertically aligned at starting position and then the inclinometer was calibrated to zero <sup>22</sup>.

Iliotibial band flexibility was measured using a modified version of the Ober's test in which an inclinometer was placed at the distal lateral thigh. In which, zero degree was recorded when thigh was horizontal, positive value was recorded if the thigh was abducted, and a negative value was recorded if the thigh was adducted past horizontal <sup>23,24</sup>.

## Functional Outcome Measures

Patient satisfaction was measured using the GROC scales, which is a commonly used method for quantifying subjects' self-perceived progress or decline over time. The GROC is scored on 15-point numerical scale from -7 to +7 where -7 represents "a very great deal worse," 0 represents "about the same" and +7 represents "a very great deal better"  $^{25}$ . An a priori score of  $\geq$ 5 was identified as the cut-off of a successful outcome  $^{25}$ . The validity and reliability of the GROC scales has been demonstrated in multiple studies  $^{26,27}$ .

The Kujala score is a 13-item self-reported questionnaire, which quantifies subjects' reported pain levels during a wide variety of activities. The scale highest scores are 100 points, which indicate lower disability. It has been shown to be a reliable and valid method for assessing functional outcomes in subjects with knee pain <sup>28,29</sup>.

The NPRS is a self-reported questionnaire with adequate reliability and validity <sup>28</sup>. Subjects were asked to rate their level of pain at baseline from three different reference points: the greatest amount of knee pain they had experienced, the least amount of knee pain they had experienced, and the level of knee pain that they were currently experiencing. These three values were then averaged to create a baseline measure of pain for each subject. All subsequent questionnaires corresponded only to subjects' present level of knee pain.

Finally, the lateral step down test (LSDT) is a measure of functionality that has been demonstrated to be both reliable and valid <sup>30</sup>. Subjects were instructed to stand with the test leg on a 15-cm step. They were then instructed to lower their body enough to cause the heel of the opposite leg to make contact with the floor directly in front of the step, and subsequently return the knee to the fully extended position. This represented a single repetition. Subjects completed as many repetitions as they could within 15 seconds, and the number of successfully completed

repetitions was recorded. This method has been widely used to ascertain functional performance in subjects with knee pain <sup>30,31</sup>.

# Statistical Analyses

A sample size of 50 subjects was estimated using a medium effect size of 0.25, a power of 0.80 and level of significance set at 0.05. However, we have complete data for 41 participants who were randomly assigned to either Protonics<sup>TM</sup> knee brace or sport cord group.

Data analysis was performed using SPSS Statistics Software version 24.0 (IBM Corp, Armonk, NY). Mean  $\pm$  SD was computed for quantitative variables and frequencies (%) for categorical variables. Normality of quantitative variables was assessed using Shapiro-Wilk test and boxplots. We compared mean age (years), Body Mass Index (kg/m²) (BMI), pain duration, and the outcome measures at baseline in both groups at baseline using independent t-test when the distribution of the variable was approximately normal and Mann-Whitney test when the distribution was not normal. The distribution of qualitative variables (gender, affected leg) by group type was examined using Chi Square test. To examine the effect of the type of intervention on outcome measures over time (baseline versus immediate versus two weeks versus four weeks), a 2x4 mixed factorial ANOVA was conducted while controlling for age at baseline since the mean age was significantly different between the two groups. The level of significance was set at  $p \le 0.05$ .

#### Results

## Subjects' Demographics

A total of 43 subjects with mean age of 28.8±5.0 years and body mass index of 25.6±4.7 kg/m<sup>2</sup> participated in the study. One subject was excluded as they had a meniscus lesion that prohibited them from participating in the study, and another subject voluntarily left the study due

to personal time constraints, therefore only data from the 41 remaining subjects who completed the prescribed intervention was analyzed. Fifty-one percent of the subjects were males (n = 21) and the majority had their right knee affected (56.1%, n=23. Twenty-one subjects (51.2%) were in the Protonics<sup>TM</sup> brace group and 20 (48.8%) in the sport cord group. There was no significant difference between the two groups in mean baseline characteristics and outcome measures at baseline except for age (30.8±5.6 vs. 26.7±3.0, p=0.01) and LSDT score (7.0±2.8 vs. 9.1±2.7, p=0.02, Table 2).

### Clinical Outcomes

Clinical improvement of subjects' patellofemoral movement impairments were assessed using four indicators: APT, hip internal/external rotation, and iliotibial band flexibility. Based on the results from all four indicators, a significant improvement was seen in all cases for both study groups for four weeks (p<0.001, Tables 3&4). APT, hip internal rotation, hip external rotation, and iliotibial band flexibility were measured at baseline, immediately following the first session, at two weeks, and at four weeks. The degree of APT decreased significantly in brace and sport cord groups (59.8% vs. 38.9%, p<0.001; respectively), however those in the brace group had sharper and quicker decrease in APT (Table 4). Hip internal rotation also increased significantly in both groups over the course of the study (p<0.001, Table 4). Similarly, hip external rotation significantly increased for both groups (p<0.001, Table 4). Lastly, iliotibial band flexibility increased significantly (p<0.001) for both the brace group and sport cord groups by 87.4% and 62.5%, respectively, with those in the brace group achieving a lower but non-significant mean score (Table 4).

### Functional Outcomes

Function of the knee joint was assessed with the Kujala Score and the lateral step-down test. Satisfaction was evaluated with the GROC, and pain was assessed according to the NPRS score. The level of satisfaction observed in the brace group was significantly higher than that of the sport cord group at the end of the four-week intervention (p<0.01, Table 3). There were no significant differences between the two groups with respect to the other three outcomes. The results of the Kujala score indicated that there was a significant improvement in knee function for both groups (13.7% vs. 10.3%, p<0.001, Table 3). The mean score for the brace group improved by 74.6%, while those in the sport cord group had 47.4% improvement. All subjects were able to perform significantly better on the lateral step test post-intervention ((p<0.001, Table 4). The brace group exhibited a 133.3% improvement in their performance, while those in the sport cord group demonstrated only an 85.3% improvement. NPRS score decreased significantly for both groups after four weeks ((p<0.001, Table 3).

# **Tables**

**Table 1. Phases of Exercise Intervention** 

| Phase | Week | Frequency | Activities |
|---|---|---|---|
| Phase I | 1 <sup>st</sup> Day of Week 1 | 1 Session | Education |
| | | | Warm-up |
| | | | Walking |
| Phase II | Weeks 1-2 | 3 Sessions per Week | Walking |
| | | | Hamstring curl in supine, prone, |
| | | | and sitting positions |
| Phase III | Weeks 3-4 | 3 Sessions per Week | Walking |
| | | | Hamstring curl in standing |
| | | | position |

Table 2. Mean  $\pm$  SD of baseline characteristics and outcome measures by study group (N=41)

| Variables | Brace (n <sub>1</sub> =21) | Sport Cord (n <sub>2</sub> =20) | p-value |
|---|---|---|---|
| Female, n (%) | 12 (57.1) | 8 (40) | 0.27 |
| Right Leg,, n (%) | 10 (47.6) | 13 (65) | 0.26 |
| Age (year) | 30.8±5.6 | 26.7±3.0 | 0.01 |
| Height ( cm) | 167.9±10.9 | 166.9±9.2 | 0.75 |
| Weight (kg) | 69.3±16.4 | 75.1±16.4 | 0.26 |
| BMI (kg/m²) | 24.4 ±4.2 | 26.8±4.8 | 0.09 |
| Pain Duration*(days) | 730 (30,4705) | 530 (37,3650) | 0.16 |
| PNRS | 4.5±1.5 | 3.8±0.7 | 0.07 |
| Kujala score | 74.8±15.0 | 79.3±8.11 | 0.24 |
| Pelvic Tilt (º) | 5.0±3.0 | 3.2±2.6 | 0.05 |
| Lateral Step-Down Test | 7.0±2.8 | 9.1±2.7 | 0.02 |
| Hip Internal Rotation | 25.9±6.3 | 28.8±7.6 | 0.19 |
| Hip External Rotation | 31.5±5.0 | 31.3±4.8 | 0.91 |
| lliotibial Band | 3.5±3.0 | 3.2±2.4 | 0.74 |

Abbreviation: SD, Standard Deviation; BMI, Body mass index

<sup>\*:</sup> median (minimum, maximum)

Table 3. Mean  $\pm$  SD of pain, global rating of change scale, and Kujala score by study group over time (N=41)

| Variable | | Protonic Bra | ace (n <sub>1</sub> =21) | | Sport Cord (n <sub>2</sub> =20) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Time | Baseline | Immediate | Two<br>Weeks | Four<br>Weeks | Baseline | Immediate | Two<br>Weeks | Four<br>Weeks | p- value over time (η²) | p-value<br>between<br>groups<br>(η²*) |
| NPRS | 4.5± 1.2 | 3.0±1.9 | 1.9±1.7 | 1.1±1.7 | 3.8±1.2 | 3.2±1.9 | 2.5±1.7 | 2.0±1.7 | <0.001<br>(0.50) | 0.9 (0.01) |
| GROC | - | 1.0±2.1 | 3.0±2.2 | 4.6±2.3 | - | 0.0±2.1 | 1.3±2.2 | 3.0±2.3 | <0.001 (0.42) | <0.01<br>(0.20) |
| Kujala<br>Score | 74.8±12.1 | - | 84.4±12.8 | 87.5±15.1 | 79.3±12.1 | - | 84.4±12.8 | 87.5±15.1 | <0.001 (0.38) | 0.39 (0.02) |

Abbreviations: PNRS, Numeric Pain Rating Scale; GROC, Global Rating of Change Scale; SD, Standard Deviation

 $<sup>^*\</sup>eta^2$  = effect size

Table 4. Comparison of mean  $\pm$  SD of HIR, HER, ITB flexibility, pelvic tilt (°), and LSDT by study group over time (N=41)

| Variable | | | Protonic Brace (n <sub>1</sub> =21) | | | Sport Cord (n <sub>2</sub> =20) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Time | Baseline | Immediate | Two<br>Weeks | Four<br>Weeks | Baseline | Immediate | Two<br>Weeks | Four<br>Weeks | p- value over time $(\eta^2)$ | p-value between group; (η²) |
| Pelvic<br>Tilt | 5.0±2.8 | 4.4±2.4 | 3.1±2.0 | 2.0±1.6 | 3.2±2.8 | 2.5±2.4 | 2.5±2.0 | 1.9±1.6 | <0.001 (0.32) | 0.08 (0.1) |
| LSDT | 7.0±2.7 | 9.6±3.3 | 13.3±3.2 | 16.3±3.3 | 9.1±2.7 | 11.8±3.3 | 14.7±3.2 | 16.8±3.3 | <0.001<br>(0.53) | 0.35 |
| HIR | 25.9±7.0 | 25.5±5.5 | 29.2±5.0 | 29.4±5.8 | 28.8±7.0 | 29.3±5.5 | 31.6±5.0 | 32.6±5.8 | <0.001 (0.24) | 0.06 (0.1) |
| HER | 31.3±4.9 | 32.2±5.0 | 32.3±5.2 | 33.9±5.7 | 31.3±4.9 | 32.2±5.0 | 32.3±5.2 | 33.9±5.7 | <0.001<br>(0.15) | 0.33 |
| ITB | 3.5±2.7 | 2.1±2.3 | 2.8±1.9 | 0.4±2.2 | 3.2±2.7 | 2.5±2.3 | 1.8±1.9 | 1.2±2.2 | <0.001 (0.23) | 0.96 (0.0) |

Abbreviations: HIR, Hip Internal Rotation; HER, Hip External Rotation; ITB, Iliotibial Band; LSDT, Lateral Step-Down Test

# **Figures**

Figure 1. Consort Flow Diagram.



**Figure 2.** Demonstration of seated hamstring curl with Protonics<sup>TM</sup> knee brace.



Figure 3. Demonstration of prone hamstring curl with sport cord.



## References

- 1. O'Connor F, et al. *Patellofemoral pain syndrome* 2018; <a href="http://www.uptodate.com/home">http://www.uptodate.com/home</a>. Accessed February 14, 2018.
- 2. Glaviano N, Kew, M, Hart, JM and Saliba, S. DEMOGRAPHIC AND EPIDEMIOLOGICAL TRENDS IN PATELLOFEMORAL PAIN. *International journal of sports physical therapy*. 2015;10(3):281-290.
- 3. Boling M, Padua, D., Marshall, S., Guskiewicz, K., Pyne, S., & Beutler, A. . Gender differences in the incidence and prevalence of patellofemoral pain syndrome. *Scandinavian Journal of Medicine & Science in Sports*. 2010;20(5):725-730.
- Surgeons AAoO. Patellofemoral pain syndrome. 2015;
   <a href="http://orthoinfo.aaos.org/topic.cfm?topic=A00680">http://orthoinfo.aaos.org/topic.cfm?topic=A00680</a>. Accessed February 14, 2018.
- 5. Lankhorst NE, Bierma-Zeinstra SM, van Middelkoop M. Risk factors for patellofemoral pain syndrome: a systematic review. *The Journal of orthopaedic and sports physical therapy*. 2012;42(2):81-94.
- 6. Witvrouw E LR, Bellemans J, Cambier D, Vanderstraeten G. . In- trinsic risk factors for the development of anterior knee pain in an athletic population: a two-year prospective study. *The American journal of sports medicine*. 2000;28:480-489.
- 7. Bogla LA ea. An update for the conservative management of patellofemoral pain syndrome: A systematic review of the literature from 2000 to 2010. *The International Journal of Sports Physical Therapy.* 2011;6:112.
- 8. Crossley K, Bennell, K., Green, S., & McConnell, J. A systematic review of physical interventions for patellofemoral pain syndrome. *Clinical Journal of Sport Medicine: Official Journal of the Canadian Academy of Sport Medicine*. 2001;11(2):103-110.
- 9. Callaghan MJ, & Selfe, J. . Patellar taping for patellofemoral pain syndrome in adults. *The Cochrane Database of Systematic Reviews*. 2012;4(CD006717).
- 10. Arroll B, Ellis-Pegler E, Edwards A, Sutcliffe G. Patellofemoral pain syndrome. A critical review of the clinical trials on nonoperative therapy. . *The American journal of sports medicine*. 1997;25(2):207-212.
- 11. Lack S, Barton, C., Vicenzino, B., & Morrissey, D. . Outcome predictors for conservative patellofemoral pain management: a systematic review and meta-analysis. . *Sports Medicine*. 2014;44(12):1703-1716.
- 12. Smith TO, Drew, B. T., Meek, T. H., & Clark, A. B. . Knee orthoses for treating patellofemoral pain syndrome. *The Cochrane Database of Systematic Reviews*. 2015;12.
- 13. Adams MA, Roughley PJ. What is intervertebral disc degeneration, and what causes it? *Spine*. 2006;31(18):2151-2161.
- 14. Denton J, Willson JD, Ballantyne BT, Davis IS. The addition of the Protonics brace system to a rehabilitation protocol to address patellofemoral joint syndrome. *The Journal of orthopaedic and sports physical therapy.* 2005;35(4):210-219.
- 15. Systems PBB. What is Protonics? 2017; <a href="https://www.protonics.info/">https://www.protonics.info/</a>. Accessed February 14, 2018.
- 16. Page P. Effectiveness of Elastic Resistance in Rehabilitation of Patients With Patellofemoral Pain Syndrome. *Sports Health*. 2011;3(2):190-194.
- 17. Khayambashi K ea. The Effects of Isolated Hip Abductor and External Rotator Muscle Strengthening on Pain, Health Status, and Hip Strength in Females With Patellofemoral Pain. *The Journal of orthopaedic and sports physical therapy.* 2012;42(1):22-29.
- 18. Denton J, Willson JD, Ballantyne BT, Davis IS. The addition of the Protonics brace system to a rehabilitation protocol to address patellofemoral joint syndrome. *Journal of Orthopaedic & Sports Physical Therapy.* 2005;35(4):210-219.

- 19. Azevedo DC, Santos H, Carneiro RL, Andrade GT. Reliability of sagittal pelvic position assessments in standing, sitting and during hip flexion using palpation meter. *J Bodyw Mov Ther*. 2014;18(2):210-214.
- 20. Herrington L. Assessment of the degree of pelvic tilt within a normal asymptomatic population. *Manual therapy.* 2011;16(6):646-648.
- 21. Han H, Kubo A, Kurosawa K, Maruichi S, Maruyama H. Hip rotation range of motion in sitting and prone positions in healthy Japanese adults. *Journal of physical therapy science*. 2015;27(2):441-445.
- 22. Cibulka MT, White DM, Woehrle J, et al. Hip pain and mobility deficits--hip osteoarthritis: clinical practice guidelines linked to the international classification of functioning, disability, and health from the orthopaedic section of the American Physical Therapy Association. *The Journal of orthopaedic and sports physical therapy.* 2009;39(4):A1-25.
- 23. Gajdosik RL, Sandler MM, Marr HL. Influence of knee positions and gender on the Ober test for length of the iliotibial band. *Clinical biomechanics (Bristol, Avon)*. 2003;18(1):77-79.
- 24. Melchione WE, Sullivan MS. Reliability of measurements obtained by use of an instrument designed to indirectly measure iliotibial band length. *The Journal of orthopaedic and sports physical therapy.* 1993;18(3):511-515.
- 25. Kamper SJ, Maher CG, Mackay G. Global Rating of Change Scales: A Review of Strengths and Weaknesses and Considerations for Design. *The Journal of Manual & Manipulative Therapy*. 2009;17(3):163-170.
- 26. Costa LO, Maher CG, Latimer J, et al. Clinimetric testing of three self-report outcome measures for low back pain patients in Brazil: which one is the best? *Spine*. 2008;33(22):2459-2463.
- 27. Farrar JT, Young JP, Jr., LaMoreaux L, Werth JL, Poole RM. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. *Pain*. 2001;94(2):149-158.
- 28. Crossley K, Bennell K, Cowan S, Green S. Analysis of outcome measures for persons with patellofemoral pain: which are reliable and valid? *Archives of physical medicine and rehabilitation*. 2004;85(5):815-822.
- 29. Paxton EW, Fithian, D. C., Stone, M. L., & Silva, P. . The reliability and validity of knee-specific and general health instruments in assessing acute patellar dislocation outcomes. *The American journal of sports medicine*. 2003;31(4):487-492.
- 30. Ross M. Test-retest reliability of the lateral step-up test in young adult healthy subjects. . *The Journal of orthopaedic and sports physical therapy.* 1997;25(2):128-132.
- 31. King A, Hancock M, Munn J. The reliability of the lateral step test. *J Sport Rehabil.* 2007;16(2):131-142.
- 32. Selhorst M, Rice W, Degenhart T, Jackowski M, Tatman M. Evaluation of a treatment algorithm for patients with patellofemoral pain syndrome: a pilot study. *International journal of sports physical therapy.* 2015;10(2):178-188.
- Hertel J, Dorfman JH, Braham RA. Lower extremity malalignments and anterior cruciate ligament injury history. *Journal of sports science & medicine*. 2004;3(4):220.
- 34. Nguyen A, Shultz, SJ. Sex differences in clinical measures of lower extremity alignment. *The Journal of orthopaedic and sports physical therapy.* 2007;37(7):389-398.
- 35. Kendall FP, McCreary EK, Provance PG. *Muscles: Testing and Function with Posture and Pain.* Lippincott Williams & Wilkins; 1999.
- 36. Earl JE, Piazza SJ, Hertel J. The Protonics Knee Brace Unloads the Quadriceps Muscles in Healthy Subjects. *Journal of Athletic Training*. 2004;39(1):44-49.
- 37. Antoun N, Kerns K, Kramer A, et al. *The Influence of the Protonics® Knee Brace on Pelvic Position.* 2002.

- 38. Jameson G, Fleisig, GS, Zheng, H, Andrews, JR, Lemak, LJ. Electromyographic responses to programmable resistance (Protonics) knee braces. The Third North American Congress on biomechanics. *Clin J Sport Med.* 1998.
- 39. Karsl G, Willet, G, Rovang, D, Miller, D. How doe the Protonics knee brace/exercise device affect knee muscle activity during functional tasks *Physical Therapy*. 1998.
- 40. Powers CM, Ward SR, Fredericson M, Guillet M, Shellock FG. Patellofemoral kinematics during weight-bearing and non-weight-bearing knee extension in persons with lateral subluxation of the patella: a preliminary study. *The Journal of orthopaedic and sports physical therapy*. 2003;33(11):677-685.
- 41. Piva S, Goodnite, EA, Childs, JD Strength Around the Hip and Flexibility of Soft Tissues in Individuals With and Without Patellofemoral Pain Syndrome. *journal of orthopaedic & sports physical therapy.* 2005;35(12).
- 42. Flack N, Nicholson, HD, Woodley, SJ. A review of the anatomy of the hip abductor muscles, gluteus medius, gluteus minimus, and tensor fascia lata. *Clin Anat.* 2012;25(6):697-708.
- 43. Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. *Annals of emergency medicine*. 1996;27(4):485-489.
- 44. Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. *Annals of emergency medicine*. 2001;38(6):633-638.
- 45. Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. *Journal of Manual & Manipulative Therapy*. 2009;17(3):163-170.
- 46. Jessee AD, Gourley MM, Valovich McLeod TC. Bracing and Taping Techniques and Patellofemoral Pain Syndrome. *Journal of Athletic Training*. 2012;47(3):358-359.
- 47. Dolak KL, Silkman C, Medina McKeon J, Hosey RG, Lattermann C, Uhl TL. Hip strengthening prior to functional exercises reduces pain sooner than quadriceps strengthening in females with patellofemoral pain syndrome: a randomized clinical trial. *The Journal of orthopaedic and sports physical therapy.* 2011;41(8):560-570.
- 48. Hoglund P. Therapeutic Exercise for Athletic Injuries. *Journal of Chiropractic Medicine*. 2003;2(2):78-79.
- 49. Logerstedt DS, Scalzitti DA, Bennell KL, et al. Knee Pain and Mobility Impairments: Meniscal and Articular Cartilage Lesions Revision 2018. *The Journal of orthopaedic and sports physical therapy.* 2018;48(2):A1-a50.